CLINICAL TRIAL: NCT05981729
Title: Feasibility of Inpatient Technology Enriched Stroke Rehabilitation During the Acute and Sub-acute Phase After Stroke
Brief Title: Technology Enriched Stroke Rehabilitation in Acute/Sub-acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Strathclyde (Other)
Collaborators: NHS Lanarkshire (Other Government)
Responsible Party: Principal Investigator, Gillian Sweeney, Principal Investigator, University of Strathclyde
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IAA_UoS/KerrBME/2023
Record Dates: First submitted 2023-07-07; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Feasibility study with convenience sample. All in patients with diagnosis of stroke and who fit criteria will be offered intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technology enhanced stroke rehabilitation (Experimental): Supported use of stroke rehabilitation technology
  Interventions: Other: Technology enriched stroke rehabilitation

INTERVENTIONS:
Other: Technology enriched stroke rehabilitation — In order to increase time spent in rehabilitation activity, participants will be prescribed and supported to use (by NHS staff) commercially available technology, such as robotics, adapted treadmills, virtual reality, and mobile digital devices such as smartphones, tablets, and wearable sensors.

SUMMARY:
Delivery of intensive rehabilitation plays an important part within stroke care and has the potential to affect rates of recovery and optimise outcomes as part of a wider multidisciplinary approach. New and innovative models of rehabilitation delivery are needed in order to bridge the gap between current staffing resources and recommended levels of rehabilitation intensity.

This study looks to investigate the feasibility and acceptability of such a model, using rehabilitation technology to enrich and enhance delivery of rehabilitation within an NHS inpatient stroke unit environment. This model of rehabilitation delivery has already been tested by the research team with community-dwelling participants in the chronic phase of stroke (over a year since stroke) and is known to be feasible and safe. Participants will be recruited from the stroke unit at University Hospital Wishaw during the acute and sub-acute phase of stroke (0-6 months since stroke), if requiring rehabilitation following a stroke and deemed medically fit enough to participate. Participants will be supported to complete activities in a newly dedicated 'technology enriched rehabilitation space' by NHS staff, in addition to their usual treatment. This will enable participants to engage in rehabilitation activities relating to their physical, cognitive, visual, communication and functional goals using equipment such as an adapted treadmill, interactive screens and tablets, upper limb exercise devices, power-assisted gym equipment and virtual reality. All devices are commercially available and known to be safe for use with stroke patients, however the use of such devices within NHS services is currently known to be under-utilised. Data will be obtained through a range of measures to monitor safety (incidence and types of adverse events), adherence (sessions/time attended, movement repetitions) and through interviews with participants, their family/carers, and staff to understand user acceptability.

DETAILED DESCRIPTION:
The Scottish Stroke Improvement Programme identifies stroke as the most common cause of severe physical disability amongst Scottish adults. Hospital care for these patients accounts for 7% of all NHS beds and 5% of the entire NHS budget. Furthermore, the number of strokes across the UK is projected to increase by 60% between 2015 and 2035.

Rehabilitation delivered by a multi-disciplinary team including Allied Health Professionals (occupational therapists [OT's], physiotherapists [PT's], and speech and language therapists [SLT's]) is known to improve functional recovery after stroke, particularly if it can be applied intensively and within enriched, stimulating environments. It is widely accepted that greater intensity, or dose, of rehabilitation improves outcomes and leads to greater and faster improvement of activities after stroke. However, a large gap exists between the minimum recommendations for stroke rehabilitation (three hours of multidisciplinary therapy a day, at least 5 days out of 7) and what the NHS are currently able to provide, given the majority of in-patient stroke units are operating below the staffing levels recommended in national clinical guidelines, and are therefore challenged to provide the amount of therapy to facilitate optimum recovery for stroke patients. An analysis of data from the UK Sentinel Stroke National Audit Programme found, on average, patients who required specific therapy following stroke received around 14 minutes of PT, 13 minutes of OT, and 7 minutes of SLT per day of inpatient stay. Therefore, new and innovative models of rehabilitation delivery are needed in order to bridge the gap between current staffing resources and recommended levels of rehabilitation intensity.

Commercially available technology, such as robotics, adapted treadmills, virtual reality, and mobile digital devices such as smartphones, tablets and wearable sensors, have been shown to be a safe and feasible method of increasing rehabilitation intensity, under the prescription and supervision of therapy staff. It can be used to enhance usual therapy and can allow stroke patients to work on physical, cognitive, visual, and communication goals, without one-to-one or 'hands on' treatment from a therapist. Despite the potential offered by rehabilitation technology to help deliver evidence-based levels of practice intensity and automated feedback without additional labour costs, currently few technologies have been adopted into everyday rehabilitation.

A well-established research group at the University of Strathclyde (UoS) Biomedical Engineering department have been developing and testing a technology-based, holistic model as a possible solution to the gap between clinical need and current provision. The technology enriched rehabilitation model has been tested under controlled conditions with chronic stroke survivors (at least one year post stroke) and shown to be feasible. While this model presents a potential method of scaling up rehabilitation delivery, and has been successfully deployed and tested for feasibility with chronic stroke, it not yet been evaluated for acute and sub-acute stroke patients or tested for clinical acceptability. This specific population has greater potential for recovery as the brain is more receptive to recovery through structural changes to neural pathways (neuroplasticity), therefore delivering higher intensity rehabilitation is therefore more critical at this phase of rehabilitation.

Recently, an NHSL occupational therapy advanced practitioner has been seconded into a research post within the UoS Biomedical Engineering department. This has created greater opportunity for collaboration between the research team at UoS and NHS Lanarkshire, to test this technology delivered rehabilitation model within an acute stroke unit where the impact of enhanced rehabilitation is likely to be greater. The Director of Hospital Services at University Hospital Wishaw (UHW) has expressed support for a technology enriched stroke rehabilitation model to be tested within the stroke unit on site and has provided a large room within the ward that can be made available for equipment (loaned from the University of Strathclyde and UK manufacturer Innerva) to be housed and used by patients under supervision from NHS staff. Funding has been secured for research assistant time from the UoS in order to support the introduction of the technology and to complete data collection. Participants will be supported to use the rehabilitation technology by trained NHS staff.

This is a mixed methods feasibility study in line with Medical Research Council recommendations for development of a complex intervention.The methodology of the study is as follows;

* Inpatients on the stroke unit, with a diagnosis of stroke, at University Hospital Wishaw, Scotland, will be assessed for eligibility by the NHS multidisciplinary team using the inclusion/exclusion criteria.
* Patients who have been identified as medically fit for rehabilitation and who fit the criteria for the study shall be highlighted to the research assistant by the NHS medical/therapy team. The researcher shall then check with the relevant members of the multi-disciplinary team that all inclusion/exclusion criteria are met before approaching the patient.
* The Participant Information Sheet and link to a supporting YouTube video with info on the study shall be supplied to the patient by the research assistant and an opportunity shall be offered for any questions from the patient and their family/carers if appropriate, with the patients consent. Informed consent shall then be taken by a University of Strathclyde research assistant only.
* Participants will be supported to access and use the rehabilitation technology, in addition to usual care, by NHS staff. This will involve the prescription of a rehabilitation technology programme by the NHS physiotherapists, occupational therapists and speech and language therapists, following usual care assessment. This is with an aim to increase rehabilitation activity within the participant's capacity, taking into account their level of impairment and fatigue. Therefore, time spent using the rehabilitation technology will be varied and tailored to meet the participant's needs. The dose and intensity of technology enriched rehabilitation will be measured and recorded, however will not be controlled for these reasons.
* The Principal Investigator (NHS occupational therapist) will hold weekly meetings with the ward therapy staff to discuss any concerns around the study or regarding participant programmes and will liaise directly with the research assistant as appropriate.
* Data collection/outcome measures will be completed as detailed in following sections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of new stroke by NHS Lanarkshire physician
* More than 48 hours since stroke event
* Deemed medically fit for rehabilitation by medical staff
* Deemed to require rehabilitation
* Able to provide informed consent

Exclusion Criteria:

* Acutely medically unwell
* Active cardiac disease, such as unstable angina
* Active delirium/significant levels of confusion
* Seizure within past 7 days
* Individual currently being managed under the Adults with Incapacity Act
* Known pregnancy
* Unable to follow verbal, written or gestured basic instructions
* Excessive pain or tonal issues which are deemed to contraindicate inclusion by medical/therapy team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of time spent on activities within the 'technology enriched rehabilitation space' | 1 year
  Time in minutes will be measured in which participants spent on activities within the 'technology enriched rehabilitation space'
Movement repetitions | 1 year
  Number of movement repetitions completed within 'technology enriched rehabilitation' sessions will be measured by use of wearable activity monitors (armbands)
Rates of recruitment and attrition | 1 year
  Percentage of eligible individual consenting to participate and percentage of people dropping/opting out before discharge.
Adherence to sessions | 1 year
  Number of sessions attended as a percentage of those available/targeted

SECONDARY OUTCOMES:
Intervention Acceptability | 1 year
  Audio-recorded semi-structured interviews will be completed with participants, family/carers and NHS staff. These interviews will be completed by a UoS research assistant. The questions posed during these interviews will focus on collecting qualitative data on the acceptability of the intervention. These shall be transcribed and thematic analysis will be used to analyse this data.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Sweeney, PhD, Principal Investigator — South Health & Social Care Partnership
Locations (1):
- University Hospital Wishaw, Wishaw, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King D, Wittenberg R, Patel A, Quayyum Z, Berdunov V, Knapp M. The future incidence, prevalence and costs of stroke in the UK. Age Ageing. 2020 Feb 27;49(2):277-282. doi: 10.1093/ageing/afz163. PMID 31957781
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100
- [Background] Gittins M, Vail A, Bowen A, Lugo-Palacios D, Paley L, Bray B, Gannon B, Tyson S. Factors influencing the amount of therapy received during inpatient stroke care: an analysis of data from the UK Sentinel Stroke National Audit Programme. Clin Rehabil. 2020 Jul;34(7):981-991. doi: 10.1177/0269215520927454. Epub 2020 Jun 7. PMID 32508132
- [Background] Kwakkel G, Kollen BJ. Predicting activities after stroke: what is clinically relevant? Int J Stroke. 2013 Jan;8(1):25-32. doi: 10.1111/j.1747-4949.2012.00967.x. PMID 23280266
- [Background] Warland A, Paraskevopoulos I, Tsekleves E, Ryan J, Nowicky A, Griscti J, Levings H, Kilbride C. The feasibility, acceptability and preliminary efficacy of a low-cost, virtual-reality based, upper-limb stroke rehabilitation device: a mixed methods study. Disabil Rehabil. 2019 Sep;41(18):2119-2134. doi: 10.1080/09638288.2018.1459881. Epub 2018 Apr 12. PMID 29644897
- [Background] Schroder J, van Criekinge T, Embrechts E, Celis X, Van Schuppen J, Truijen S, Saeys W. Combining the benefits of tele-rehabilitation and virtual reality-based balance training: a systematic review on feasibility and effectiveness. Disabil Rehabil Assist Technol. 2019 Jan;14(1):2-11. doi: 10.1080/17483107.2018.1503738. Epub 2018 Oct 14. PMID 30318952
- [Background] Kerr A, Smith M, Reid L, Baillie L. Adoption of Stroke Rehabilitation Technologies by the User Community: Qualitative Study. JMIR Rehabil Assist Technol. 2018 Aug 17;5(2):e15. doi: 10.2196/rehab.9219. PMID 30120086
- [Background] Kerr A, Keogh M, Slachetka M, Grealy M, Rowe P. An Intensive Exercise Program Using a Technology-Enriched Rehabilitation Gym for the Recovery of Function in People With Chronic Stroke: Usability Study. JMIR Rehabil Assist Technol. 2023 Jul 21;10:e46619. doi: 10.2196/46619. PMID 37477954
- [Background] National Clinical Guideline for Stroke for the UK and Ireland, 2023 edition. Royal College of Physicians, London UK.
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508